CLINICAL TRIAL: NCT02354417
Title: A Phase 1 Trial of a Single ProHema® CB Product (Ex Vivo Modulated Human Cord Blood Cells) Following Myeloablative Conditioning for Pediatric Patients With Hematologic Malignancies
Brief Title: A Phase 1 Trial of a Single ProHema® CB Product for Pediatric Patients With Hematologic Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Fate Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FT1050-04
Record Dates: First submitted 2014-09-25; First posted 2015-02-03 (Estimated); Results first posted 2018-10-10 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-02

CONDITIONS: Hematologic Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ProHema-CB (Experimental): All subjects will receive treatment with ProHema-CB (ex-vivo modulated human cord blood cells) transplant.
  ProHema-CB (the prostaglandin derivative, 16,16-dimethyl prostaglandin E2 also referred to as FT1050) will be prepared and administered in one of two formulations, based upon subject weight:
  For subjects > 35 kg, ProHema-CB will be administered as 150 mL product in a blood bag via gravity infusion. It will be infused at 10 mL to 15 mL per minute, for a total infusion time of 10 to 15 min.
  For subject's ≤ 35 kg, ProHema-CB will be administered as a 50 mL product in a syringe via syringe pump.o It will be infused at 5 mL/kg per hour for a total infusion time of up to ~1 hour.
  Interventions: Biological: Biological: ProHema-CB

INTERVENTIONS:
Biological: Biological: ProHema-CB — Each subject will receive one administration of ProHema-CB unit transplant.

SUMMARY:
This is an open-label, safety study of a single ProHema-CB product administered following myeloablative conditioning regimen in pediatric subjects with hematologic malignancies.

DETAILED DESCRIPTION:
A maximum of 18 eligible male and female subjects (1 to 18 years old, inclusive) will be enrolled and treated in the trial at approximately 3 to 5 centers within the U.S. These 18 subjects will consist of 3 cohorts of 6 subjects each. The cohorts will be defined by age: 1 to 4 years; > 4 to 12 years; and > 12 to 18 years. These cohorts will be enrolled simultaneously.

All subjects will be admitted to the hospital, per institutional practice, and will receive a myeloablative conditioning regimen, after which they will receive an HLA-matched or partially matched ProHema-CB unit on study Day 0.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged 1 to 18 years, inclusive.
2. Subjects with hematologic malignancies for whom allogeneic stem cell transplantation is deemed clinically appropriate.

   1. Acute Myelogenous Leukemia (AML) in high risk 1st or subsequent CR
   2. Acute Lymphoblastic Leukemia (ALL) in CR
   3. NK cell lymphoblastic leukemia in any CR
   4. Biphenotypic or undifferentiated leukemia in 1st or subsequent CR
   5. Myelodysplastic Syndrome (MDS) at any stage.
   6. Chronic Myelogenous Leukemia (CML) All subjects with evidence of CNS leukemia must be treated and be in CNS CR to be eligible for trial.
3. Lack of 5-6/6 HLA matched related or 8/8 HLA A, B, C, DRß1 matched unrelated donor; or unrelated donor not available within appropriate timeframe, as determined by the transplant physician.
4. Availability of suitable primary and secondary umbilical cord blood (UCB) units.
5. Adequate performance status, defined as:

   1. Subjects ≥ 16 years: Karnofsky score ≥ 70%.
   2. Subjects < 16 years: Lansky score ≥ 70%.
6. Cardiac: Left ventricular ejection fraction at rest must be > 40%, or shortening fraction > 26%.
7. Pulmonary:

   1. Subjects > 10 years: DLCO (diffusion capacity) > 50% of predicted (corrected for hemoglobin)
   2. FEV1, FVC > 50% of predicted; Note: If unable to perform pulmonary tests, then O2 saturation > 92% on room air.
8. Renal: Serum creatinine within normal range for age, or if serum creatinine outside normal range for age, then renal function (creatinine clearance or GFR) > 70mL/min/1.73m2.
9. Hepatic: Bilirubin ≤ 2.5 mg/dL (except in the case of Gilbert's syndrome or ongoing hemolytic anemia); and ALT, AST and Alkaline Phosphatase ≤ 5 × ULN.
10. Signed IRB approved Informed Consent Form (ICF).

Exclusion Criteria:

1. Female subjects that are pregnant or breastfeeding.
2. Evidence of HIV infection or HIV positive serology.
3. Current uncontrolled bacterial, viral or fungal infection.
4. Prior allogeneic hematopoietic stem cell transplant.
5. Autologous transplant < 12 months prior to enrollment.
6. Prior autologous transplant for the disease for which the UCB transplant is being performed.
7. Active malignancy other than the one for which the UCB transplant is being performed within 12 months of enrollment.
8. Inability to receive TBI.
9. Requirement of supplemental oxygen.
10. HLA-matched related donor able to donate.
11. Use of an investigational drug within 30 days prior to screening.
12. Subject is unlikely to comply with the protocol requirements, instructions and study-related restrictions

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2014-12; Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Storgard, MD, Study Director — Fate Therapeutics
Locations (2):
- United States (2):
  - City of Hope, Duarte, California
  - Boston Children's Hospital, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Groups:
- ProHema-CB: All subjects will receive treatment with ProHema-CB (ex-vivo modulated human cord blood cells) transplant.
  ProHema-CB (the prostaglandin derivative, 16,16-dimethyl prostaglandin E2 also referred to as FT1050) will be prepared and administered in one of two formulations, based upon subject weight:
  For subjects > 35 kg, ProHema-CB will be administered as 150 mL product in a blood bag via gravity infusion. It will be infused at 10 mL to 15 mL per minute, for a total infusion time of 10 to 15 min.
  For subject's ≤ 35 kg, ProHema-CB will be administered as a 50 mL product in a syringe via syringe pump.o It will be infused at 5 mL/kg per hour for a total infusion time of up to ~1 hour.
  Biological: ProHema-CB: Each subject will receive o
Period: Overall Study
Arm/Group | ProHema-CB
Started | 3
Completed | 2
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- ProHema-CB: All subjects will receive treatment with ProHema-CB (ex-vivo modulated human cord blood cells) transplant.
  ProHema-CB (the prostaglandin derivative, 16,16-dimethyl prostaglandin E2 also referred to as FT1050) will be prepared and administered in one of two formulations, based upon subject weight:
  For subjects > 35 kg, ProHema-CB will be administered as 150 mL product in a blood bag via gravity infusion. It will be infused at 10 mL to 15 mL per minute, for a total infusion time of 10 to 15 min.
  For subject's ≤ 35 kg, ProHema-CB will be administered as a 50 mL product in a syringe via syringe pump.o It will be infused at 5 mL/kg per hour for a total infusion time of up to ~1 hour.
  Biological: ProHema-CB: Each subject will receive one administration of ProHema-CB unit transplant.
Arm/Group | ProHema-CB
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: Years] | 15.7 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 1
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 3
Weight (kg) [Mean (Standard Deviation); unit: kg] | 73.4 (28.8)

OUTCOME MEASURES:

1. Primary Outcome: Safety Profile, Primarily Assessed by Neutrophil Engraftment
Description: To describe the safety profile of ProHema-CB after myeloablative conditioning in pediatric patients with hematologic malignancies. The safety profile will primarily be assessed by neutrophil engraftment.
Time Frame: Neutrophil engraftment by Day 42
Measure: Count of Participants; unit: Participants
Arm/Group | ProHema-CB
Number analyzed (Participants) | 3
Participants | 3

ADVERSE EVENTS:
Time Frame: During the First Year of Transplant
Description: Serious Adverse Events and Adverse Events assessed as possibly or probably related to ProHema are included below.
Arm/Group | ProHema-CB
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ProHema-CB (N=3)
Mucosal inflammation (General disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes